CLINICAL TRIAL: NCT05924555
Title: Exercise Intolerance Study in Long Chain Fatty Acid Oxidation Disorders
Acronym: EXCITE LcFAOD
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Stichting Stofwisselkracht (Unknown)
Responsible Party: Principal Investigator, Dr. Mirjam Langeveld, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL83869.018.23
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Long-chain Fatty Acid Oxidation Disorders
Keywords: Long-chain Fatty Acid Oxidation disorders; Exercise intolerance; Cardiopulmonary exercise test
MeSH Terms: interventions — Hand Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LcFAOD-patients: Patients with long-chain Fatty Acid Oxidation including CPT2-, CACT-, VLCAD-, LCHAD-, or MTP-deficiency
  Interventions: Other: Intermittent cardiopulmonary exercise test; Other: Incremental cardiopulmonary exercise test; Other: Echography of upper leg; Other: Hand grip strength with hand dynamometer; Other: Fill in questionnaires regarding physical activity
- Healthy controls: Controls are matched based on Age, Sex, BMI and comparable activity score assessed using the SQUASH questionnaire
  Interventions: Other: Intermittent cardiopulmonary exercise test; Other: Incremental cardiopulmonary exercise test; Other: Echography of upper leg; Other: Hand grip strength with hand dynamometer; Other: Fill in questionnaires regarding physical activity

INTERVENTIONS:
Other: Intermittent cardiopulmonary exercise test — Exercise test with step-change from rest to a relatively low constant workload.
Other: Incremental cardiopulmonary exercise test — Exercise test with incremental workload until maximal workload.
Other: Echography of upper leg — Determine upper leg muscle size
Other: Hand grip strength with hand dynamometer — Determine muscle strength
Other: Fill in questionnaires regarding physical activity — SQUASH, mMRC, questionnaire designed to report myopathic symptoms in LcFAOD patients.

SUMMARY:
In this study, the exercise tolerance in patients with long-chain fatty acid oxidation disorders (LcFAOD) will be compared to that of healthy volunteers who are carefully matched in terms of age, sex, BMI and physical activity score. The study aims to assess exercise capacity using cardiopulmonary exercise (CPX) tests and activity monitoring over a 7-day period. The hypothesis of the study is that LcFAOD patients will exhibit greater oxygen debt during short periods of exercise compared to healthy individuals. These findings will contribute to a better understanding of exercise intolerance in LcFAOD patients and may guide the development of targeted interventions, such as exercise training programs and enable the analysis of effectiveness of (new) treatments.

DETAILED DESCRIPTION:
Background:Long-chain fatty acid oxidation disorders (LcFAOD) are a group of autosomal recessive disorders that impair the utilization of long-chain fatty acids as an energy source. Exercise intolerance is a commonly reported symptom in adult patients with LcFAOD, but its severity varies significantly among individuals. In addition, little is currently known about the natural progression of exercise intolerance in this group of patients, and reliable outcome measures to assess treatment efficacy remain scarce. In this study, we will evaluate the exercise capacity in LcFAOD patients using intermittent CPX, and determine whether this yields outcome parameters that can be used to determine the course of exercise intolerance over the patients lifetime and evaluate treatment effectiveness.

Hypothesis: Exercise intolerance in LcFAOD patients will be reflected in differences in VO2/VCO2 and heart rate kinetics during short periods of exercise compared to healthy subjects.

Primary Objective: 1. Objectify and quantify exercise intolerance in LcFAOD patients. 2. Determine the relationship between the measured exercise intolerance and patient-reported symptoms, daily life functioning, as well as known markers of disease severity.

Secondary Objective(s): 3. Determine the aetiology of exercise intolerance in LcFAODs. 4. Determine whether the intermittent exercise protocol can be used to establish the course of exercise intolerance and provide clinical outcome measure for future intervention studies.

Methods: Participants will be asked to wear an activity monitor (Activ8) for a period of 7 days. The participants will also perform two cardiopulmonary exercise (CPX) tests (one intermittent and one incremental). During the CPX tests gas exchange, ventilation, blood pressure and cardiac output will be measured and exhaustion level monitored. Blood samples will be taken before the first and after the second CPX test. The grip strength (Maximal Voluntary Contraction) and the leg muscle size (echography) will be assessed. Body composition (using BIA) will be assessed.

Approximately a year later all procedures, including the wearing of the activity monitor, will be repeated in all patients. Some participants will be asked to perform the two exercise tests again within two weeks of their first visit. This way reproducibility of the intermittent exercise protocol can be tested.

ELIGIBILITY:
Inclusion Criteria:

* LC-FAOD patients:
* Men and women (age ≥18 years) with a confirmed diagnosis of carnitine palmitoyltransferase 2 (CPT2) deficiency, Carnitine-acylcarnitine translocase (CACT) deficiency, Mitochondrial Trifunctional protein (MTP) deficiency, Very-long-chain acyl-CoA dehydrogenase (VLCAD) deficiency or Long-chain 3-hydroxyacyl-CoA dehydrogenase (LCHAD) deficiency.

Healthy control subjects:

- Healthy men and women age ≥ 18 years

Exclusion Criteria:

LcFAOD patients:

* Pregnancy
* Recent acute myocardial infarction (<6 months prior to inclusion)
* Uncontrolled arrhythmia/severe conduction disorder causing hemodynamic compromise
* Implantable pacemaker or other cardiac device with complete ventricular pacing
* Uncontrolled heart failure with hemodynamic compromise
* Uncontrolled hypertension (Systolic Blood Pressure >150 mmHg and Diastolic Blood Pressure >100 mmHg on repeated measurements)
* Active infection, anemia, severe renal dysfunction (estimated Glomerular filtration rate < 30 ml/min/1,73m2), or other chronic disease likely to significantly impact exercise performance
* History of severe asthma or chronic obstructive pulmonary disease
* Active use of medication likely to affect exercise tolerance

Healthy controls:

* All abovementioned exclusion criteria for LcFOAD patients
* History of smoking - History of asthma, chronic obstructive pulmonary disease, heart failure, heart surgery, heart rhythm disorders or congenital heart diseases
* Chronic illness (including orthopedic, endocrinological, hematological, malignant, gastrointestinal, neurological, muscle or inflammatory disorders) likely to significantly impact on exercise performance
* > 6 alcohol units per day or > 14 alcohol units per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients with long chain fatty acid oxidation disorders are under follow-up are eligible to participate in the study. Each patients will be compared to a matched healthy control subject (one healthy subject can serve as a control for more than one LcFAOD patient). Matching will be done by age (± 3 years), sex, BMI (± 2 kg/m2) and a comparable activity score assessed using a questionnaire (the Short Questionnaire to Asses Health enhancing physical activity (SQUASH).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
1. Differences in V'O2/ V'CO2/heart rate kinetics during the intermittent exercise test between LcFAOD patients and healthy control subjects | At rest (baseline) and during the intermittent CPX test (30 min)
Anaerobic threshold (ml/kg/min) | During maximum exercise (max 30 min).
  Pulmonary involvement/Cardiac dysfunction/Skeletal muscle alterations
Ventilation reserve (L) | During maximum exercise (max 30 min).
  Pulmonary involvement/Skeletal muscle alterations
CO2 ventilation equivalent (L/L) | During maximum exercise (max 30 min).
  Pulmonary involvement/Cardiac dysfunction
Cardiac Output (L/min) | During maximum exercise (max 30 min).
  Cardiac dysfunction
Heart rate reserve (per minute) | During maximum exercise (max 30 min).
  Cardiac dysfunction
Muscle size on echography (cm) | Baseline
  Skeletal muscle alterations
Muscle strength via resistance test (kg) | Baseline
  Skeletal muscle alterations

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Langeveld, MD PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No